CLINICAL TRIAL: NCT05854680
Title: To Investigate the Metabolomics in the Subjects With Long Term Tai Chi Chuan Practice
Status: Completed | Type: Observational
Sponsor: Sheng-Teng Huang (Other)
Responsible Party: Sponsor-Investigator, Sheng-Teng Huang, Attending physician, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Other Study IDs: CHUH108-REC2-020
Record Dates: First submitted 2023-04-19; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Tai Chi Chuan; Metabolomics
Keywords: Traditional Chinese medicine; Yin and Yang; Tai Chi Chuan; Metabolomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Long term: Tai Chi has been practiced for at least five years, regular practice, at least three times a week, each practice for at least 30 minutes.
- Short term: Tai Chi practice time is less than three months, regular practice, at least three times a week, each practice for at least 30 minutes.

SUMMARY:
The new biomedical technology including genomics and metabolomics will be applied to the subjects with TCC practice to investigate clinical symptoms and signs expression. The investigators will compare the related molecular pathways especially focusing on immune and inflammation between long term practice and beginner groups.

DETAILED DESCRIPTION:
Tai Chi has been developed and spread in the eastern Asia, even the whole world for a long time. It is an exercise to coordinate mind, breathing and body movements slowly and continuously. Tai Chi is regarded as a good and useful sport to strengthen the body. In recent ten years, more and more evidence demonstrated the benefits of Tai Chi especially by meta-analysis studies. These studies revealed that Tai Chi can lower blood pressure, including systolic and diastolic blood pressure, fasting blood glucose, HbA1c, total cholesterol, triglyceride and low-density lipoprotein cholesterol, as well as preventing bone mineral density (BMD) loss in special populations. Tai Chi also helps the patients with Parkinson's disease reduce falls due to improving balance and functional mobility, and improve the symptoms of depression and anxiety. Recently, people are currently facing how to reduce the risk factors of cardiovascular diseases, promote physical and mental health and strengthen muscles and bones, and so on. Regarding the role of Tai Chi in immunity, Tai Chi is helpful to improve immune function, however, the results are still inconsistent that it needs to be elucidated.

Metabolomics technology is widely used in the fields of medicine and life sciences. Through mass spectrometry analysis, quantitative and qualitative changes in biomarkers can be used to identify biochemical metabolic pathways or effects that might be involved. The number of studies on metabolomics applications has grown rapidly over the past decade, however, little has been done to examine the physiological effects of Tai Chi practice. In addition, with the advancement of science and technology, the sensitivity and measurement method of the mass spectrometer have been improved, which is more suitable for understanding the physiological changes by Tai Chi exercises. After all, the exact cellular molecular mechanisms remain largely unknown after the practice of Tai Chi.

In order to understand the health care of Tai Chi, the investigators designed this clinical control study to observe its clinical benefits from both traditional Chinese medicine and Western medicine. The investigators mainly compared long-term Tai Chi practitioners with beginner by TCM diagnosis and physical analysis to identify the differences and changes in TCM syndromes. At the same time, modern medical-related molecular biotechnology is used to detect changes in immunity and metabolomics analysis. Based on the views from macro to micro, it may provide important clues for clinical trials of related diseases with application of Tai Chi exercise in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women aged over 20 and under 65.
2. Participants agreed to join the trial by fully understanding the purpose of the study and the entire trial process and then signed an informed consent.

Exclusion Criteria:

1. Age of subjects was under 20 or more than 65 years old.
2. Subjects were using immunosuppressive or chemotherapy drugs.
3. With a history of drug abuse.
4. Pregnant or breastfeeding women.
5. Mental or behavioral abnormalities such as schizophrenia, depression, suicidal ideation, etc.
6. Suffering from serious diseases such as myocardial infarction, heart failure, arrhythmia, chronic respiratory obstructive diseases, cancers, gastrointestinal bleeding (OB positive), etc.
7. Subjects with abnormal blood count, abnormal liver function (>2 times the normal value), and abnormal renal function.
8. Subjects were still participating in other clinical trials.
9. Subjects were not willing sign the informed consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The enrolled normal subjects were confirmed by the Tai Chi Association and the research PI. The long-term group has practiced Tai Chi for at least five years, and the short-term group has been practiced for less than three months. Men and women aged between 20 and 65 are included. We collected all of subjects' basic information, four diagnosis associated with TCM Syndrome Differentiation, FACIT-Fatigue scale, PSQI, BDI-II, SF-36 questionnaire scale, blood tests for CBC, liver and kidney function as well as metabolite analysis.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Serum metabolites | on the day of admission.
  Collect blood and measure the level of serum metabolites .
Plasma Cytokines | on the day of admission.
  Collect blood and measure the level of plasma cytokines. Comparison of cytokine values between different groups.
Constitution in Chinese Medicine Questionnaire (CCMQ) | completed on the day of admission.

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale (Version 4) | completed on the day of admission.
  uses 13 short fatigue-related questions to measure an individual level of fatigue in daily life over the past week. Each rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). The scores for each item are summed to obtain a total score ranging from 0 to 52. A score of less than 30 indicates severe fatigue, and a higher score indicates less fatigue.
36-Item Short Form Health Survey (SF-36) | completed on the day of admission.
  contains eight domains: physical functioning, physical health problems, bodily pain, general health perceptions, vitality, social functioning, emotional problems, and mental health. This is scored on a scale ranging from 0 to 100, with higher scores indicating better health-related quality of life.
Pittsburgh Sleep Quality Index (PSQI) | completed on the day of admission.
  uses a self-administered questionnaire and fills in 19 items to evaluate sleep quality in the previous month
BDI-II score | completed on the day of admission.
  consists of 21 sets of questions, each of which is self-administered with a score ranging from 0 to 3. Ultimately, a total score of 0-13 is considered minimal, 14-19 mild, 20-28 moderate, and 29-63 severe

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Teng Huang, MD PhD, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: No